CLINICAL TRIAL: NCT03938948
Title: The Efficacy of Visible Red Light for Promoting the Growth of Human Scalp Hair for Both Male and Female - An Open-label Study
Brief Title: Low Level Light Therapy (LLLT) for Hair Growth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Awareable Technologies Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COH02.01
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Male Pattern Baldness; Female Pattern Baldness
MeSH Terms: conditions — Alopecia | interventions — Phototherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treatment Arm (Experimental): 62 participants shall be enrolled
  Interventions: Device: low-level laser/light therapy

INTERVENTIONS:
Device: low-level laser/light therapy — Participants will wear light therapy devices for 14 weeks

SUMMARY:
A total of 62 participants will receive red light (660 nm) to the scalp through a specially designed light therapy device integrated into a conventional hat. Each treatment will be 30 min per session applied on every other day for 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between the ages of 18 and 60 years
* Diagnosed AGA in the past 12 months for male (Fitzpatrick I-IV, Hamilton-Norwood IIa-V ) and female (Fitzpatrick I-IV, and Ludwig-Savin Baldness Scale I-2, I-3, I-4, II-1, II-2 baldness patterns)

Exclusion Criteria:

* Known Photosensitivity
* Using any oral or topical substance for hair growth
* Having Tattoo, hair transplantation, scalp reduction, malignancy or hair weave in the scalp are with alopecia
* Known medical conditions that could negatively affect hair growth, such as infections, connective tissue disease
* Currently or plan to be on a calorie-restricted diet during study participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2019-04-11 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Hair Density | 14 weeks
  Individual participant's hair density will be measured at the end of 14 weeks and compared with the baseline density measure at the start of the treatment.
Hair Density | 14 weeks
  Mean hair density for the participants after 14 weeks will be compiled and compared with the mean density of the participants' at the start of the study to determine changes.

SECONDARY OUTCOMES:
Hair Follicle Change | 14 weeks
  Both individual and all participants' follicles shall be analyzed to determine the percent of change in hair follicle anagen/telogen ratio

CONTACTS AND LOCATIONS:
Overall Officials: Michael Will, MD, Principal Investigator
Locations (1):
- Will Surgical Arts, Ijamsville, Maryland, United States